CLINICAL TRIAL: NCT02280668
Title: Investigating Muscle Repair in Response to Icing Therapy Post Eccentric Muscle Damage Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Christopher Chekay, Undergraduate Student, Wilfrid Laurier University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4177
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Muscle Damage
Keywords: muscle; muscle repair; tissue repair; eccentric exercise; force loss; icing; cold therapy; DOMS; soreness; recovery
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Active Comparator): Will perform the eccentric muscle damage exercise and will not perform any icing interventions post damage. These participants will be the control group.
  Interventions: Other: the eccentric muscle damage exercise
- Icing Protocol 1 (Experimental): Will perform the eccentric muscle damage exercise and will begin the icing intervention immediately after the muscle damage. The icing protocol will be icing the elbow flexor muscles for 10 minutes with a cold pack followed by 10 minutes with no icing and another 10 minutes of elbow flexor muscle icing. The participants will perform this protocol every day at approximately the same time for the duration of the study.
  Interventions: Other: Icing Therapy; Other: the eccentric muscle damage exercise
- Icing Protocol 2 (Experimental): Will perform the eccentric muscle damage exercise and will begin the icing intervention 6 hours post muscle damage. The icing protocol will be icing the elbow flexor muscles for 10 minutes with a cold pack followed by 10 minutes with no icing and another 10 minutes of elbow flexor muscle icing. The participants will perform this protocol every day at approximately the same time for the duration of the study.
  Interventions: Other: Icing Therapy; Other: the eccentric muscle damage exercise

INTERVENTIONS:
Other: Icing Therapy — Participants will be randomly assigned into 3 experimental groups. Icing Protocol 1 has participants apply cold packs under the supervision of the principal investigators to their elbow flexor region for 10 minutes on, 10 minutes off, followed by an additional 10 minutes on, starting at time 0. Icing Protocol 2 follows the same procedure but it begins 6 hours after the participant has completed their eccentric muscle damaging exercise and is to be done at home without the supervision of the principal investigators. Both protocols require the participants to repeat their icing procedures every 24 hours until their involvement with the study is finished, which is 7 days in duration. The third experimental group is the control group and will not participate in an icing therapy during the duration of the study.
  Other Names: Cold Therapy; Cryotherapy
  Arms: Icing Protocol 1; Icing Protocol 2
Other: the eccentric muscle damage exercise

SUMMARY:
The purpose of our research is to investigate the effects of applying cold therapy, or "icing," to injured muscles in terms of strength recovery and muscle soreness amelioration following unaccustomed exercise.

DETAILED DESCRIPTION:
The objective is to determine whether or not injured muscles that are subject to icing after eccentrically damaging exercise recover their strength quicker and/or have less muscle soreness than those that do not receive any icing treatment after damaging exercise and if any differences in effectiveness between two icing protocols exist. Baseline measures of peak torque of the dominant arm's elbow flexor muscles will be measured by concentric and isometric contractions prior to participants undergoing eccentric muscle damaging exercise. Participants will be randomly assigned into 3 different experimental groups of approximately 15 participants each. The first group will begin "Icing Protocol 1" at time 0 (or as close to). The second group will begin "Icing Protocol 2" six hours after their initial eccentric muscle damaging exercise. The remaining group will not receive any icing treatment; they are the control group. Participants will be brought back into the lab at specific post-exercise times (0h, 24h, 48h, 96h, and 7 days) to complete peak torque measures as they did with baseline measures prior to eccentric muscle damage. Measures of delayed onset muscle soreness (DOMS) will also be taken at baseline and during scheduled follow up times for participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy students attending Wilfrid Laurier University with no previous history of upper body muscle damage and live in close proximity to the University so they can attend all lab sessions. Ideally they have not performed any upper body resistance training within the last 4 months.

Exclusion Criteria:

* Previous history of muscle, joint, or ligament injuries in the surrounding area of their dominant are elbow flexor region.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Peak torque strength measures determined using the CYBEX-NORM Testing and Rehabilitation System | Within 7 days post eccentric muscle damage
Delayed onset muscle soreness determined using the VAS scale of perceived muscle soreness | Within 7 days post eccentric muscle damage

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tiidus, PhD, Study Director — Wilfrid Laurier University, Faculty of Health Sciences
Locations (1):
- Wilfrid Laurier University, Waterloo, Ontario, Canada